CLINICAL TRIAL: NCT00124800
Title: The Effect of Tinnitus Retraining Therapy on Subjective and Objective Measures of Chronic Tinnitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tinnitus Research Consortium (Other)
Responsible Party: Carol Bauer, Professor of Otolaryngology, SIU School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-014
Record Dates: First submitted 2005-07-27; First posted 2005-07-28 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Tinnitus
Keywords: tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Behavioral: Tinnitus retraining therapy — Sound therapy and counseling
Device: Sound therapy — sound therapy and counselling

SUMMARY:
The objective of this study is to examine the efficacy of tinnitus retraining therapy (TRT) as a treatment of chronic tinnitus in people with limited hearing loss. The study design is prospective, randomized, double-blind, with repeated measures. The null hypothesis states there will be no difference in subjective measures of tinnitus severity between subjects treated with standard TRT and subjects treated with sham TRT.

DETAILED DESCRIPTION:
The specific aims of the study are to:

* Evaluate the efficacy of TRT in reducing the objective magnitude of tinnitus.
* Evaluate the efficacy of TRT in reducing the subjective awareness and impact of tinnitus.
* Determine the therapeutic time course of improvement in tinnitus.
* Determine the long-term improvement in tinnitus derived from TRT.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-pulsatile tinnitus

Exclusion Criteria:

* Hyperacusis
* Subjective hearing loss
* Objective hearing loss with pure tone average greater than 35 dB sound pressure level (SPL)
* Evidence of significant depression or suicidal ideation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change in objective measure of tinnitus loudness using psychoacoustic matching task | 18 months
Change in subjective handicap rating of tinnitus using a standardized questionnaire | 18 months

SECONDARY OUTCOMES:
Change in subjective ratings of tinnitus loudness, annoyance and awareness | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Bauer, MD, Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

REFERENCES:
- See also: Related Info — http://siumed.edu/surgery